CLINICAL TRIAL: NCT06621901
Title: Effect of High Protein Diet on Endoplasmic Reticulum Stress
Brief Title: Effect of Protein on Endoplasmic Reticulum Stress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Aslı Onur Canaydın, Research Assistant of Department of Nutrition and Dietetics, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ERU-BD-AOC-03
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Effect of High Protein Diet on Endoplasmic Reticulum Stress
Keywords: Endoplasmic reticulum stress; High protein diet; Oxidative stress
MeSH Terms: interventions — Diet, High-Protein

STUDY DESIGN:
Intervention Model Description: It consists of two parallel groups receiving a high-protein diet and a normal-protein diet.
Who Masked: Participant
Masking Description: The content of the diet will be given to the participants without specifying it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Protein Diet (Experimental): The energy composition of the high protein diet will be calculated as 40% carbohydrate, 30% protein and 30% fat. It will be stated that individuals should not eat anything other than the foods to be sent during the weeks of the diet.
  Interventions: Other: High Protein Diet
- Normal Protein Diet (Experimental): The energy composition of the high protein diet will be calculated as 55% carbohydrate, 15% protein and 30% fat. It will be stated that individuals should not eat anything other than the foods to be sent during the weeks of the diet.
  Interventions: Other: Normal Protein Diet

INTERVENTIONS:
Other: High Protein Diet — Individuals will be placed on a high protein diet for 10 days.
  Arms: High Protein Diet
Other: Normal Protein Diet — Individuals will be placed on a normal protein diet for 10 days.
  Arms: Normal Protein Diet

SUMMARY:
This study was planned to provide information about the effect of short-term high protein diet (HPD) feeding on endoplasmic reticulum stress. The definition of HPDs cannot be determined exactly. They are defined differently by various scientific authorities. However, the target is for protein to be approximately 30% of total energy in HPD. It has been determined that HPDs increase satiety, thermogenesis, and provide body weight loss and maintenance of loss. In general, there is evidence that HPDs provide more body weight loss in a short time compared to low protein diets. It has been emphasized that the effect of high protein diet on weight loss is related to creating satiety, thus reducing food intake and increasing thermogenesis. However, the physiological, biochemical and molecular events that occur due to HPD feeding are not fully understood and the results have not been explained. It has been determined that the effects of HPDs last between 1 and 6 days and 6 months. The absence of any study in the literature on the short-term and long-term effects of HPD on oxidative events in humans reveals the original value of this study. Therefore, considering that long-term HPD feeding may increase the risk of cardiovascular disease, blood pressure and blood lipid levels, the effect of short-term HPD feeding on endoplasmic reticulum stress will be investigated in order to avoid these side effects. Blood analyses planned for this prospective analytical study will be performed in GENKÖK Laboratory. Healthy individuals will be administered 10 days of HPD and a 10-day normal diet as a control.

DETAILED DESCRIPTION:
Today, many people are trying various nutritional models/diets to reduce body weight. One of the most popular of these diets is the diets that reduce carbohydrate intake. Western societies generally avoid high carbohydrate and fat intake. For this reason, interest in high protein intake in diets is increasing day by day. Although there is no general consensus on what a high protein diet (HPD) is, HPD applied for weight loss is a diet that contains approximately 30% of the energy provided by protein. The World Health Organization (WHO) has defined obesity as an endemic public problem and stated that its prevalence is increasing. With the increase in obesity, individuals are trying various dietary changes to achieve weight loss. These include diets with more regular macro and micronutrient patterns such as the Mediterranean Diet and DASH diet, and diets that may cause deficiencies in terms of macro and micronutrients such as Atkins, South Beach, Zone and Stillman, which contain high protein. The most important reasons for the interest in HPD are that it causes rapid weight loss and provides a feeling of satiety. This positive effect of HPDs on weight loss has attracted the attention of dietitians and has led them to increase the protein ratio in diets.

It is known that HPDs provide more effective results in body weight loss compared to low-protein diets. It is suggested that this effect occurs as a result of increased thermogenesis, increased satiety and suppressed appetite, and decreased glycemic index and glycemic load due to the replacement of refined carbohydrates with proteins. In addition to this positive effect on weight loss, HPD nutrition also has possible short- and long-term side effects. Known complications of long-term HPD nutrition include increased risk of cardiovascular disease, blood pressure, blood lipids, and renal dysfunction. Cardiovascular problems in particular are a source of concern, as they will eliminate the short-term positive effect of HPD on weight loss and increase the burden of cardiovascular disease in the long term. Studies generally focus on HPD and weight loss; there is limited data on the relationship between HPD nutrition and metabolic dysfunction such as endothelial dysfunction, inflammatory markers, antioxidant status, and other chronic diseases. The physiological, biochemical and molecular events that occur due to high protein diets are not fully understood and their results have not been explained.

High protein diets (especially low carbohydrate diets) are thought to have negative effects because they cause a decrease in fruit and vegetable consumption. In those who eat HPD, especially those with insufficient vitamins A, C and E in their diets, this will have a negative effect on antioxidant systems and will lead to the development of many chronic and metabolic diseases in the long term. Despite the positive effects of HPD applied as a weight loss diet in the short term, it is thought that the oxidative stress and inflammation it will create in the long term will cause an increase in chronic and metabolic diseases and comorbidities. This increase in the disease burden will increase health expenditures both individually and socially.

Increasing evidence has shown that ROS and inflammation increase the production of reactive oxygen species (ROS). There is a direct link between ROS production and cellular events such as protein oxidation and protein folding. ROS and ROS production are integral components of ERS and are not merely consequences of ERS induction. It has been reported that increased ERS triggers ERS and can cause various types of cell death. First, some forms of ROS can disrupt ER protein folding and trigger ERS. Exogenous oxidants such as ROS producers, peroxides, metal ions, and lipid oxidation products can activate some aspects of the UPR. 7-ketocholesterol, a major oxidation product of cholesterol in atherosclerotic plaque, induces the UPR in macrophages and vascular smooth muscle cells. The 7-ketocholesterol-activated UPR is suppressed by the antioxidant N-acetylcysteine, indicating that ERS induction is dependent on ERS. However, other forms of ROS such as hydrophene peroxide (H2O2) can only stimulate mild or specific components of the UPR. A study has determined that selenocysteine-free phospholipid hydroperoxide GPx (NPGPx), a member of the glutathione peroxidase (GPx) family, senses OS in the ER lumen and then forms a disulfide bond with GRP78, resulting in chaperone activity. Furthermore, OS induced during protein misfolding in the ER has led eukaryotic cells to develop antioxidative stress responses to restore cellular redox homeostasis. The PERK branch of the UPR induces two transcription factors, ATF4 and Nrf2, that transactivate antioxidative stress response genes, including SODs, HO-1, glutathione transferase, and uncoupler mitochondrial protein 2. The PERK signaling pathway of the UPR acts to maintain redox balance during ERS through activation of ATF4 and Nrf2. Small molecular antioxidants such as butylated hydroxyanisole (BHA) can prevent ERS-induced apoptosis and promote proper protein folding and secretion, suggesting a critical role for ERS in protein misfolding. As another example, two mitochondrial-targeted antioxidants, Mitoquinone and MitoTempol, have been shown to reduce mitochondrial ERS, ERS, and cell death in β cells. Antioxidants can suppress both ERS and ERS. Therefore, treatments targeting both stressors may be effective in preventing both ERS and metabolic, neurodegenerative, immune, and neoplastic diseases.

Therefore, the aim of this planned study is to examine the effect of HPD, which has gained popularity especially with its increasing use in weight loss diets, on ERS. Thus, scientific literature will be produced that can prevent the possible negative effects of HPD and at the same time, it can support the reduction of ERS, which is effective in the course of various chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Being between 19-45 years of age,
* Not changing physical activity throughout the study,
* Having a BMI of 18.5-24.9 kg/m2,
* Being healthy

Exclusion Criteria:

* Having a BMI of <18.5 and ≥25 kg/m2,
* Having a chronic disease,
* Smoking and drinking alcohol,
* Using vitamin-mineral supplements and herbal supplements,
* Being pregnant or breastfeeding,
* Having entered menopause,
* Being on any diet.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Endoplasmic reticulum stress after high protein diet | Day after diet end
  After the diet, endoplasmic reticulum stress parameters (GRP78, PERK, Nrf2 and GPx-1) will be measured in the blood.

IPD SHARING:
Plan to Share IPD: No